CLINICAL TRIAL: NCT00533767
Title: Prospective Follow Up of Household Contacts and Hantavirus Transmission Study Among Index and Additional Cases in Chile
Brief Title: Hantavirus Transmission in Households in Chile
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and was inadvertently added to the system.
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07-0013
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Hantavirus Infections
Keywords: Hantavirus cardiopulmonary syndrome, Andes virus, Chile
MeSH Terms: conditions — Hantavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to evaluate the transmission of hantavirus in Chile. It is an observational study that will look at close household contacts of people who have been diagnosed with hantavirus infections that result in a serious illness to see how frequently they become infected. Subjects who enroll in the study will donate samples of body fluids (e.g., blood, saliva, stool, urine, respiratory and vaginal secretions) to allow the researchers to see if hantavirus is present in those fluids and if so, how much. Subjects will also be interviewed to identify household conditions that may be associated with transmission. Up to 76 index cases (people who are first diagnosed with hantavirus cadiopulmonary illness) and up to 140 of their close contacts will be enrolled. Subjects will be followed for about 6 weeks.

DETAILED DESCRIPTION:
Hantavirus cardiopulmonary syndrome (HCPS) has a case fatality rate of 40-50 percent. Andes virus (ANDV) is the primary pathogen in Chile and Argentina. This is a prospective observational study to access the incidence of and risk factors associated with transmission of HCPS to close household contacts from HCPS index cases including examination of the shedding of virus in various body fluids as a factor in transmissibility. The study will enroll 76 cardiopulmonary syndrome HCPS index cases and 140 of their close household contacts, age 2 and older, at risk for contracting HCPS.

The index cases will participate for the initial visit; the household contact participants will be followed for 35 days. The primary objectives of this study are: to estimate the secondary attack rate of hantavirus infection among close household contacts of an HCPS case after one incubation period of follow up; to use personal interviews and questionnaires to assess and compare risk activities and demographic factors in close household contacts who develop HCPS with those contacts who do not identify specific high-risk activities such as exposure to saliva or respiratory secretions; to use personal interviews and questionnaires to assess and compare risk activities and demographic factors in index cases (the first case in the household) versus household contacts who do not develop HCPS; and to determine the prevalence of hantavirus in various body fluids in index patients with HCPS and in household contacts who acquire infection and consequently determine any association of presence of virus in a body fluid with phase of infection.

Both infectious virus (culture) and viral genomic RNA (quantitative RT-PCR) will be measured. The secondary objectives of this study will be: to determine the quantity of hantavirus in various body fluids in index patients with HCPS and in household contacts that acquire infection and consequently determine any association of presence of virus in a body fluid with phase of infection. Both infectious virus (culture) and viral genomic RNA (quantitative RT-PCR) will be measured; to develop a predictive statistical model where the epidemiological and the virological variables (cultures, ANDV antibodies, PCR, neutralizing antibodies, HSV 1 and 2 antibodies) could be scored and used to predict a new case within a household group; to determine the feasibility of rapid viral diagnostic testing to determine whether virologic results can be obtained sufficiently in advance of the onset of illness to permit more effective triage of patients who are indeed about to develop HCPS; and to determine the sequences of ANDV from index and additional cases to establish the extent of sequence identity from viruses within and outside of family clusters.

The primary endpoints of this study are: to determine the incidence of additional cases of hantavirus (ANDV) among close household contacts of a confirmed index case during a complete incubation period of follow up; evaluate risk activities and demographic factors associated with increased risk of transmission of ANDV between index cases and members of households and their respective index cases; measure risk activities and demographic factors associated with increased risk of acquisition of ANDV from environmental sources by comparing index cases with household contacts that do and do not develop HCPS; and determine the presence of virus and measure of viral RNA in body fluids over time in index cases and in additional cases in household contacts.

The secondary endpoints will be: to determine the most sensitive culture approach for detection of ANDV in body fluids at different stages of infection; identify the best model to predict the occurrence of an additional case within a family group; evaluate nucleotide similarity as ancillary marker to enrich or de-enrich the probability of person to person transmission of AND virus. The duration of this study is expected to be 3 years.

ELIGIBILITY:
Inclusion Criteria:

Index Cases:

1. Confirmed diagnosis, positive hantavirus IgM assay or detection of hantavirus in plasma or serum by RT-PCR.
2. Signed informed consent form.
3. Less than 96 hours have transpired since the diagnosis was confirmed.

Household Contact

1. Any person, 2 years of age or older, who has been in close contact with the index case at any point from 30 days before to 7 days after the onset of symptoms in the index case.
2. Close contact must include: sexual contact and/or deep kissing and/or slept in same bed and/or provided direct care to index case.

Exclusion Criteria:

Index Cases

1. Index case does not have or agree to give the names of his/her close contacts.
2. Not a suitable candidate in the opinion of the investigator.

Household Contact

1. Confirmed current or previous infection with Andes virus.
2. Younger than 2 years of age.
3. Unavailable for follow up or not a suitable candidate in the opinion of the investigator.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 76 index cases with hantavirus cardiopulmonary syndrome and their close household contacts
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Estimate the secondary attack rate among close household contacts of index cases with hantavirus cardiopulmonary syndrome in Chile | 35 days

SECONDARY OUTCOMES:
Determine the quantity of hantavirus in bodily fluids in persons with hantavirus infection | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Mertz, MD, Principal Investigator — University of New Mexico
Locations (1):
- Universidad Catolica de Chile, Santiago, Chile